CLINICAL TRIAL: NCT01843972
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Oral Doses of BI 691751 in Healthy Male Volunteers in a Randomised, Single-blind, Placebo-controlled Design (Part I) and Investigation of Relative Bioavailability of BI 691751 Given as Tablet and Oral Solution to Healthy Male Subjects in an Open, Randomised, Single-dose, Single Period Parallel Group Design (Part II).
Brief Title: Safety of Single Rising Doses and Relative Bioavailability of BI 691751
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1334.1; 2012-005721-67 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

ARMS (10):
- BI 691751 dose 2 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751 dose 3 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751 dose 4 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751 dose 5 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751 dose 6 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751 dose 7 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- BI 691751dose 1 (part I) (Experimental): single dose given as oral solution
  Interventions: Drug: BI 691751
- Placebo (part I) (Placebo Comparator): placebo solution
  Interventions: Drug: Placebo
- BI 691751 tablet (part II) (Experimental): single dose given as 1 tablet
  Interventions: Drug: BI 691751
- BI 691751 solution (part II) (Active Comparator): single dose given as oral solution
  Interventions: Drug: BI 691751

INTERVENTIONS:
Drug: BI 691751 — oral solution BI 691751, dose 6
  Arms: BI 691751 dose 6 (part I)
Drug: BI 691751 — oral solution
  Arms: BI 691751 solution (part II)
Drug: Placebo — placebo solution
  Arms: Placebo (part I)
Drug: BI 691751 — oral solution BI 691751, dose 2
  Arms: BI 691751 dose 2 (part I)
Drug: BI 691751 — oral solution BI 691751, dose 5
  Arms: BI 691751 dose 5 (part I)
Drug: BI 691751 — 1 tablet
  Arms: BI 691751 tablet (part II)
Drug: BI 691751 — oral solution BI 691751, dose 3
  Arms: BI 691751 dose 3 (part I)
Drug: BI 691751 — oral solution BI 69175, dose 4
  Arms: BI 691751 dose 4 (part I)
Drug: BI 691751 — oral solution BI 691751, dose 7
  Arms: BI 691751 dose 7 (part I)
Drug: BI 691751 — oral solution BI 69175, dose 1
  Arms: BI 691751dose 1 (part I)

SUMMARY:
To investigate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of single rising doses of BI 691751 in healthy male subjects (part I).

To investigate the relative bioavailability of BI 691751 given as tablet versus oral solution (part II)

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. Subjects must be able to understand and comply with study requirements
3. Age from 18 to 55 years
4. BMI range: from 18.5 to 29.9 kg/m2
5. Known genotype as specified in the study protocol

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1334.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- BI 691751 Dose 1 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 69175, dose 1 (0.5 mg powder)
- BI 691751 Dose 2 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 691751, dose 2 (1.5 mg powder)
- BI 691751 Dose 3 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 691751, dose 3 (5 mg powder)
- BI 691751 Dose 4 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 69175, dose 4 (15 mg powder)
- BI 691751 Dose 5 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 691751, dose 5 (30 mg powder)
- BI 691751 Dose 6 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 691751, dose 6 (60 mg powder)
- BI 691751 Dose 7 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 691751, dose 7 (90 mg powder)
- BI 691751 Tablet (Part II): single dose given as 1 tablet
  BI 691751: 1 tablet (10 mg)
- BI 691751 Solution (Part II); Extensive Metabolizers: single dose given as oral solution BI 691751: oral solution (10 mg)
  5 subjects had no measurable concentration of BI 691751 because a drug-free solution has been administered by mistake. Therefore their results were excluded from all analyses.
Period: Overall Study
Arm/Group | Placebo (Part I) | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Tablet (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers
Started | 13 | 6 | 5 | 6 | 6 | 6 | 5 | 5 | 17 | 12
Completed | 13 | 6 | 5 | 6 | 5 | 6 | 5 | 5 | 17 | 12
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): includes all subjects who were documented to have taken at least 1 dose of study medication.
Groups:
- BI 691751dose 1 (Part I): single dose given as oral solution
  BI 691751: oral solution BI 69175, dose 1 (0.5 mg powder)
- Total: Total of all reporting groups
Arm/Group | Placebo (Part I) | BI 691751dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Tablet (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers | Total
Number analyzed (Participants) | 13 | 6 | 5 | 6 | 6 | 6 | 5 | 5 | 17 | 12 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (8.2) | 31.2 (8.0) | 32.0 (8.4) | 34.5 (6.8) | 26.5 (5.2) | 37.5 (6.0) | 29.2 (2.6) | 30.2 (8.0) | 32.2 (9.3) | 35.8 (10.2) | 31.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 13 | 6 | 5 | 6 | 6 | 6 | 5 | 5 | 17 | 12 | 81

OUTCOME MEASURES:

1. Primary Outcome: AUC0-72h (Part II)
Description: AUC0-72h (area under the concentration-time curve of the analyte of BI 691751 in plasma over the time interval from 0 to 72 h) (part II).
  PPS-BA included all subjects in the TS who were randomised to the BA part, who provided at least one observation for at least one primary endpoint, had no important protocol violations relevant for the statistical evaluation of BA and did not experience emesis at or before twice the median tmax.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h and 72h after drug administration
Population: Per protocol set for evaluation of bioavailability (PPS-BA). Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- BI 691751 Tablet Extensive Metabolizers (Part II): single dose given as 1 tablet; extensive metabolizers;
  BI 691751: 1 tablet (10 mg)
- BI 691751 Tablet Poor Metabolizers (Part II): single dose given as 1 tablet; poor metabolizers;
  BI 691751: 1 tablet (10 mg)
Arm/Group | BI 691751 Tablet Extensive Metabolizers (Part II) | BI 691751 Tablet Poor Metabolizers (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 12 | 5 | 7
nmol*h/L | 2740 (26.1) | 3050 (20.5) | 2800 (22.2)
Statistical Analysis 1: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Solution (Part II); Extensive Metabolizers; Only extensive CYP2D6 metabolisers were selected: 12 (all) subjects of group 'BI 691751 tablet extensive metabolizers (part II)' and 7 (all investigated) subjects of group 'BI 691751 solution (part II) '; Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 97.88, 90% CI 2-sided [79.963 to 119.809], Standard Deviation 24.8 — The geometric mean ratio is calculated as the geometric mean of 'BI 691751 tablet extensive metabolizers (part II)' divided by the geometric mean of 'BI 691751 solution (part II)'
Statistical Analysis 2: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Tablet Poor Metabolizers (Part II); Comparison of poor metabolisers (5 (all) subjects of group 'BI 691751 tablet poor metabolizers (part II)') and extensive metabolisers (12 (all) subjects of group 'BI 691751 tablet extensive metabolizers (part II)'); Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 111.20, 90% CI 2-sided [88.596 to 139.576], Standard Deviation 24.7 — The geometric mean ratio was calculated as the geometric mean of the poor metabolisers divided by the geometric mean of the extensive metabolisers

2. Primary Outcome: Cmax (Part II)
Description: Cmax (maximum measured concentration of the analyte of BI 691751 in plasma) (part II)
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug administration
Population: PPS-BA. Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 691751 Tablet Extensive Metabolizers (Part II) | BI 691751 Tablet Poor Metabolizers (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 12 | 5 | 7
nmol/L | 223 (33.6) | 207 (31.3) | 220 (14.4)
Statistical Analysis 1: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Solution (Part II); Extensive Metabolizers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 101.31, 90% CI 2-sided [80.593 to 127.351], Standard Deviation 28.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Tablet Poor Metabolizers (Part II); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 92.69, 90% CI 2-sided [68.662 to 125.119], Standard Deviation 33.0 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Cmax (Part I)
Description: Cmax (maximum measured concentration of BI 691751 in plasma) (part I)
  Time frame:
  Dose 1 and 2: 1 hour (h) before drug administration (admin) and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h and 168h after drug admin
  Dose 3 and 4: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h (dose group 4 only), 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h and 240h after drug admin
  Dose 5 to 7: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 336h, 432h, 528h, 624h and 720h after drug admin
  Dose 8: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug admin
Time Frame: for dose 1 & 2: up to 168h, for dose 3 & 4: up to 240h, for dose 5 to 8: up to 720h
Population: Per protocol set for evaluation of dose proportionality (PPS-DP): This subject set includes all subjects of the TS who were randomised to active treatment in the single rising dose part or BA part, and had no important PVs relevant for the statistical evaluation of dose proportionality. Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 5 | 5 | 7
nmol/L | 3.45 (15.5) | 18.3 (39.3) | 88.9 (59.1) | 729 (21.5) | 1320 (31.5) | 3320 (46.7) | 4180 (22.2) | 220 (14.4)
Statistical Analysis 1: Comparison: BI 691751 Dose 4 (Part I) vs BI 691751 Dose 5 (Part I) vs BI 691751 Dose 6 (Part I) vs BI 691751 Dose 7 (Part I); Test type: Non-Inferiority or Equivalence — This was non-confirmatory testing; Regression, Linear; Slope = 1.0233, 95% CI 2-sided [0.8265 to 1.2201]

4. Secondary Outcome: AUC0-infinity (Part I)
Description: AUC0-infinity (area under the concentration-time curve of BI 691751 in plasma over the time interval from 0 extrapolated to infinity) (part I)
  Time frame:
  Dose 1 and 2: 1 hour (h) before drug administration (admin) and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h and 168h after drug admin
  Dose 3 and 4: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h (dose group 4 only), 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h and 240h after drug admin
  Dose 5 to 7: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 336h, 432h, 528h, 624h and 720h after drug admin
  Dose 8: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug admin
Time Frame: for dose 1 & 2: up to 168 hours (h), for dose 3 & 4: up to 240h, for dose 5 to 8: up to 720h
Population: PPS-DP. Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 0 | 0 | 6 | 5 | 6 | 5 | 5 | 7
nmol*h/L |  |  | 1140 (34.5) | 7250 (15.9) | 11900 (27.2) | 24500 (20.0) | 41000 (26.9) | 3630 (28.5)
Statistical Analysis 1: Comparison: BI 691751 Dose 4 (Part I) vs BI 691751 Dose 5 (Part I) vs BI 691751 Dose 6 (Part I) vs BI 691751 Dose 7 (Part I); Dose proportionality of BI 691751 was explored using a power model (regression model applied to log-transformed data); Test type: Non-Inferiority or Equivalence — This was non-confirmatory testing; Regression, Linear; Slope = 0.9686, 95% CI 2-sided [0.8107 to 1.1266]

5. Secondary Outcome: AUC0-tz
Description: AUC0-tz (area under the concentration-time curve of BI 691751 in plasma over the time interval from 0 up to the last quantifiable data point) (Part I and Part II)
  Time frame:
  Dose 1 and 2: 1 hour (h) before drug administration (admin) and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h and 168h after drug admin
  Dose 3 and 4: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h (dose group 4 only), 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h and 240h after drug admin
  Dose 5 to 7: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 336h, 432h, 528h, 624h and 720h after drug admin
  Dose 8: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug admin
Time Frame: Part 1: for dose 1 & 2: up to 168 hours (h), for dose 3 & 4: up to 240h, for dose 5 to 7: up to 720h; Part 2: up to 720h
Population: PPS-DP for part I and PPS-BA for part II. Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Tablet Extensive Metabolizers (Part II) | BI 691751 Tablet Poor Metabolizers (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 0 | 5 | 6 | 6 | 6 | 5 | 5 | 12 | 5 | 7
nmol*h/L |  | 29.5 (18.4) | 791 (45.4) | 6310 (15.4) | 11400 (28.3) | 24100 (21.1) | 40500 (27.2) | 3150 (32.0) | 3460 (17.4) | 3300 (28.5)
Statistical Analysis 1: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Solution (Part II); Extensive Metabolizers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 95.48, 90% CI 2-sided [74.414 to 122.511], Standard Deviation 30.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 691751 Tablet Extensive Metabolizers (Part II) vs BI 691751 Tablet Poor Metabolizers (Part II); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANOVA; Geometric mean ratio (net) = 109.80, 90% CI 2-sided [84.376 to 142.894], Standard Deviation 28.8 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: BI 691751 Dose 4 (Part I) vs BI 691751 Dose 5 (Part I) vs BI 691751 Dose 6 (Part I) vs BI 691751 Dose 7 (Part I); Test type: Non-Inferiority or Equivalence — This was non-confirmatory testing; Regression, Linear; Slope = 1.0312, 95% CI 2-sided [0.833 to 1.1790]

6. Secondary Outcome: t1/2 (Part I)
Description: t1/2 (terminal half-life of the analyte of BI 691751 in plasma) (part I)
  Time frame:
  Dose 1 and 2: 1 hour (h) before drug administration (admin) and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h and 168h after drug admin
  Dose 3 and 4: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h (dose group 4 only), 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h and 240h after drug admin
  Dose 5 to 7: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 336h, 432h, 528h, 624h and 720h after drug admin
  Dose 8: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug admin
Time Frame: for dose 1 & 2: up to 168 hours (h), for dose 3 & 4: up to 240h, for dose 5 to 8: up to 720h
Population: Pharmacokinetic (PK) set (PKS) which includes all subjects of the treated set were were randomised to active treatment in the single rising dose part of bioavailability part, and had no important protocol violations relevant for the statistical evaluation of further PK parameters. Only subjects with calculable PK parameter were analysed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 0 | 0 | 6 | 5 | 6 | 5 | 5 | 7
h |  |  | 65.4 (37.8) | 97.4 (63.3) | 74.9 (49.2) | 57.2 (34.3) | 78.3 (16.9) | 59.4 (57.1)

7. Secondary Outcome: Tmax (Part I)
Description: tmax (time from dosing to maximum measured concentration of BI 691751) (part I)
  Time frame:
  Dose 1 and 2: 1 hour (h) before drug administration (admin) and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h and 168h after drug admin
  Dose 3 and 4: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h (dose group 4 only), 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h and 240h after drug admin
  Dose 5 to 7: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 336h, 432h, 528h, 624h and 720h after drug admin
  Dose 8: 1h before drug admin and 20 min, 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 144h, 216h, 384h, 552h and 720h after drug admin
Time Frame: for dose 1 & 2: up to 168 hours (h), for dose 3 & 4: up to 240h, for dose 5 to 8: up to 720h
Population: PKS
Measure: Median (Full Range); unit: h
Arm/Group | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Solution (Part II); Extensive Metabolizers
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 5 | 5 | 7
h | 0.667 [0.333 to 0.667] | 0.667 [0.350 to 0.667] | 0.842 [0.333 to 2.02] | 0.500 [0.333 to 0.667] | 0.350 [0.333 to 0.667] | 0.667 [0.333 to 1.50] | 0.667 [0.333 to 1.02] | 0.667 [0.333 to 1.50]

8. Primary Outcome: Frequency of Subjects With Drug-related Adverse Events (Part I)
Description: Frequency of subjects with drug-related Adverse Events (AEs) (Part I)
Time Frame: Part I: 'Day1 to Day21 for Dose 1, 2,3 &4 and Day1 to Day45 for Dose group 5,6 & 7
Population: Treated Set (TS): all subjects who were documented to have taken at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo (Part I) | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I)
Number analyzed (Participants) | 13 | 6 | 5 | 6 | 6 | 6 | 5 | 5
Participants | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day1 to Day21 for Dose group 1, 2,3 & 4 and Day1 to Day45 for Dose group 5,6 & 7. Part II: Day1 to Day 45.
Description: Subjects randomised to 0.5 mg sol. or 1.5 mg sol. were planned by the CTP to be observed for 8 to 21 days, subjects randomised to 5 mg sol. or 15 mg sol. for 11 to 21 days, and subjects randomised to 10 mg sol., 10 mg tab., 30 mg sol., 60 mg sol., or 90 mg sol. for 31 to 45 days after treatment.
Arm/Group | Placebo (Part I) | BI 691751 Dose 1 (Part I) | BI 691751 Dose 2 (Part I) | BI 691751 Dose 3 (Part I) | BI 691751 Dose 4 (Part I) | BI 691751 Dose 5 (Part I) | BI 691751 Dose 6 (Part I) | BI 691751 Dose 7 (Part I) | BI 691751 Tablet (Part II) | BI 691751 Solution (Part II); Extensive Metabolizers
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/17 | 1/12
Other Adverse Events (participants affected / at risk) | 5/13 | 1/6 | 2/5 | 2/6 | 2/6 | 1/6 | 3/5 | 4/5 | 5/17 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part I) (N=13) | BI 691751 Dose 1 (Part I) (N=6) | BI 691751 Dose 2 (Part I) (N=5) | BI 691751 Dose 3 (Part I) (N=6) | BI 691751 Dose 4 (Part I) (N=6) | BI 691751 Dose 5 (Part I) (N=6) | BI 691751 Dose 6 (Part I) (N=5) | BI 691751 Dose 7 (Part I) (N=5) | BI 691751 Tablet (Part II) (N=17) | BI 691751 Solution (Part II); Extensive Metabolizers (N=12)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part I) (N=13) | BI 691751 Dose 1 (Part I) (N=6) | BI 691751 Dose 2 (Part I) (N=5) | BI 691751 Dose 3 (Part I) (N=6) | BI 691751 Dose 4 (Part I) (N=6) | BI 691751 Dose 5 (Part I) (N=6) | BI 691751 Dose 6 (Part I) (N=5) | BI 691751 Dose 7 (Part I) (N=5) | BI 691751 Tablet (Part II) (N=17) | BI 691751 Solution (Part II); Extensive Metabolizers (N=12)
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.